CLINICAL TRIAL: NCT06431490
Title: A Study to Evaluate the Efficacy, Safety, and Immunogenicity of TQB2102 for Injection in the Treatment of HER2-positive Locally Advanced or Metastatic Biliary Tract Cancer
Brief Title: A Study of TQB2102 for Injection in the Treatment of HER2-positive Biliary Tract Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-Ib/II-01
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2102 for injection (Experimental): Intravenous infusion, administered every 3 weeks, 21 days as a treatment cycle, 6/8 cycles.
  Interventions: Drug: TQB2102 for injection

INTERVENTIONS:
Drug: TQB2102 for injection — TQB2102 for injection is a HER2 dual-antibody-drug Conjugate (ADC)

SUMMARY:
To evaluate the efficacy and safety TQB2102 for injection in the treatment of patients with Her2-positive biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ age ≤75 years; Eastern Cooperative Oncology Group (ECOG) score 0 to 1;
* Test subjects with HER2 expression or amplification or mutation require immunohistochemistry of HER2 3+ or HER2 2 and positive for in situ hybridization (ISH);
* The main organs function well;
* Meet the criteria for advanced biliary tract cancer:

  1. Biliary tract carcinoma confirmed by histology or cytology;
  2. Non-operable locally advanced, recurrent and/or metastatic disease with at least one measurable lesion according to Evaluation criteria for the efficacy of solid tumors (RECIST) 1.1 criteria;
  3. Failure of previous standard treatment.
* Women of reproductive age should agree that effective contraception must be used during the study period and for 6 months after the end of the study, and that serum or urine pregnancy tests are negative within 7 days prior to study enrollment; Men should agree that effective birth control must be used during the study period and for 6 months after the end of the study period;
* The subjects voluntarily joined the study, signed the informed consent, and the compliance was good.

Exclusion Criteria:

* Complicated diseases and medical history:

  1. Have had or are currently suffering from other malignant tumors within 3 years before the first medication;
  2. Unmitigated toxic effects higher than grade 1 of Common Terminology Criteria for Adverse Events (CTCAE) due to any previous treatment;
  3. Major surgical treatment, significant traumatic injury, or long-term unhealed wounds or fractures have been received within 4 weeks prior to initial medication;
  4. Patients with any bleeding or bleeding events ≥CTCAE grade 3 within 4 weeks before the first dose; Aortic/venous thrombosis events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism, occurred within 6 months prior to initial administration; Treatment with low molecular weight heparin was permitted and antiplatelet drugs were prohibited throughout the study period;
  5. Active viral hepatitis with poor control;
  6. There is a history of active tuberculosis, idiopathic pulmonary fibrosis, institutional pneumonia, drug-induced pneumonia, radiation pneumonia requiring treatment or active pneumonia with clinical symptoms;
  7. Have a history of psychotropic drug abuse and can not quit or have mental disorders;
  8. People who are ready to undergo or have previously received allogeneic bone marrow transplantation or solid organ transplantation;
  9. Have a history of hepatic encephalopathy;
  10. Currently on or recently used (within 7 days before the start of study treatment) aspirin (>325 mg/ day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel, and cilostazol;
  11. Subjects with any severe and/or uncontrolled disease.
* Tumor related and treatment:

  1. For subjects who have received chemotherapy, immunotherapy within 3 weeks before the first dose, radiation therapy or small molecule targeted drugs within 2 weeks, or who are still within the 5 half-lives of the drug (as the shortest time of occurrence), the washout period is calculated from the end time of the last treatment;
  2. Within 2 weeks before the first use of the drug, the treatment of Chinese patent drugs with anti-tumor indications specified in the National Medical Products Administration (NMPA) approved drug instructions;
  3. Imaging including computed tomography (CT) or magnetic resonance imaging (MRI) shows that the tumor has invaded important blood vessels, or the investigator determines that the tumor is highly likely to invade important blood vessels during the follow-up study period and cause fatal massive bleeding;
  4. Uncontrolled pleural effusion, pericardial effusion or moderate to severe ascites that still require repeated drainage;
  5. Obvious biliary obstruction (except for total bilirubin ≤ 2× upper limit of normal (ULN) after endoscopic stent placement and percutaneous transhepatic biliary drainage);
  6. Known spinal cord compression, cancerous meningitis, with symptoms of brain metastases, or symptoms controlled for less than 4 weeks.
* Research treatment related:

  1. Known allergy to study drug excipients;
  2. Have previously received anti-HER2 therapy drugs (only for the second stage, the first stage is not limited);
  3. Patients who require immunosuppressive, systemic, or absorbable topical hormone therapy for immunosuppressive purposes and who continue to use it for 7 days prior to initial administration (except for corticosteroids <10 mg per day of prednisone or other therapeutic hormones).
  4. Participants who participated in and used other anti-tumor clinical trials within 4 weeks before the first medication.
  5. According to the judgment of the researcher, there is a situation that seriously endangers the safety of the subjects or affects the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AE) and serious adverse events (SAE) | From the time the subject signed the informed consent until 28 days after the last dose/start of the new antitumor therapy
  Any adverse medical event that occurred from the time the subject signed the informed consent until 28 days after the last dose/start of the new antitumor therapy (whichever came first).
Phase II Recommended Dose (RP2D) | Baseline up to 24 weeks
  Phase II Recommended Dose (RP2D)

SECONDARY OUTCOMES:
Objective response rate (ORR) | Baseline up to 36 weeks
  The percentage of subjects achieving complete response (CR) or partial response (PR) as assessed by the investigator based on the Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
Progression-free survival (PFS) | Baseline up to 36 weeks
  The time between first medication and first disease progression or death from any cause.
Disease control rate (DCR) | Baseline up to 36 weeks
  The first assessment was complete response, partial response, and time to disease stabilization.
Disease response time (DOR) | Baseline up to 36 weeks
  First assessed as complete or partial response to first disease progression or time of death from all causes.
Overall survival (OS) | Baseline up to 36 weeks
  Time from first use to death from any cause

CONTACTS AND LOCATIONS:
Locations (43):
- China (43):
  - Fuyang Cancer Hospital, Fuyang, Anhui
  - Anhui Second People's Hospital, Hefei, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Tsinghua Changgeng Hospital, Beijing, Beijing, Beijing Municipality
  - First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Gansu Provincial Tumor Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Guangxi University Affiliated Hospital, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - AnYang Tumor Hospital, Anyang, Henan
  - Luoyang Central Hospital (Zhengzhou University Affiliated Luoyang Central Hospital), Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan University Zhongnan Hospital, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Dongtai People'S Hospital, Yancheng, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Chifeng City Hospital, Chifeng, Neimengu
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Cancer Hospital of Shan dong First Medical University, Jinan, Shandong
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Seventh People's Hospital, Shanghai, Shanghai Municipality
  - The Third Affiliated Hospital of PLA Navy Medical University, Shanghai, Shanghai Municipality
  - First Hospital of Shangxi Medical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang University Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang